CLINICAL TRIAL: NCT02872467
Title: Prenatal Cocaine, Nasal Oxytocin, and Maternal Psychophysiology
Acronym: NOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-3053
Record Dates: First submitted 2016-07-12; First posted 2016-08-19 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2022-02

CONDITIONS: Substance Abuse Problem; Pregnancy
Keywords: Cocaine; Mothers; Pregnant women; Postpartum women; Oxytocin; Substance use disorders; Substance abuse; Prenatal substance use; stress
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Syntocinon treatment (Experimental): Syntocinon spray, 24 IU twice daily (A single dose will be delivered consisting of 6 intranasal insufflations (3 in each nostril) which is equivalent to a total of 24 international units (IU) of oxytocin twice daily).
  Interventions: Drug: Syntocinon treatment
- Placebo (Placebo Comparator): Placebo nasal spray vials will contain the same ingredients in the nasal preparation, but without oxytocin.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Syntocinon treatment — 24 IU twice daily (A single dose will be delivered consisting of 6 intranasal insufflations (3 in each nostril) which is equivalent to a total of 24 international units (IU) of oxytocin twice daily).
  Other Names: Nasal Oxytocin treatment
  Arms: Syntocinon treatment
Other: Placebo — Placebo nasal spray vials will contain the same ingredients in the nasal preparation, but without oxytocin.
  Arms: Placebo

SUMMARY:
The purpose of this research is to study the effects of nasal oxytocin administration on maternal behaviors that may be influenced by cocaine use during pregnancy. 32 mothers with prenatal use of cocaine during the current pregnancy will be studied at 3-6 months postpartum, when they will complete 3 study visits, a 2-week double-blind trial of twice daily nasal spray (oxytocin or placebo) and 4 telephone interviews. All information collected is confidential.

DETAILED DESCRIPTION:
Participation for mothers when they are 3-6 months postpartum includes:

* Visit 1: Questionnaires and interviews about participants' health, pregnancy, moods, psychological history and drug use during pregnancy and postpartum.
* Visit 2: Pregnancy & drug tests (results are confidential), blood samples and vital signs, video-taped mother-infant interaction, speech task, instruction re: using nasal spray (oxytocin or placebo) & self-administration of first nasal spray dose, followed by 90 minutes of monitoring.
* At-home nasal spray: Twice daily (before breakfast and supper) nasal spray self-administration for 14 days.
* Visit 3: Pregnancy & drug tests (results are confidential), blood samples and vital signs, video-taped mother-infant interaction, speech task, interviews and questionnaires about mothers' experience with the nasal spray, and changes in mood or physical discomfort during the 2-weeks when taking the nasal spray.
* 3 telephone interviews while subjects are taking nasal spray, and 1 post-trail telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 3-6 months postpartum at start of testing
* Cocaine use during current pregnancy (by self-report or medical record of prenatal urine toxicology)
* Exclusive Formula-feeding for all infant milk feedings (no infant feeds will be breast milk)
* Healthy singleton pregnancy
* English fluency that will allow informed consent

Exclusion Criteria:

* Pregnancy or plans to become pregnant during participation in the study
* Not using effective birth control methods to prevent pregnancy
* Breastfeeding for any infant milk feedings
* Mother is not currently living with the infant during the trial period
* Multiple birth (twin, triplet or greater)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-05; Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
The effects of a 2-week trial of twice nasal oxytocin compared with placebo on maternal sensitivity | 2 weeks

SECONDARY OUTCOMES:
The effects of a 2-week trial of nasal oxytocin compared with placebo on maternal reactivity to a social stressor indexed by change in vascular resistance from pre- to post-test nasal spray. | 2 weeks
The effects of a 2-week trial of nasal oxytocin compared with placebo on maternal reactivity to a social stressor indexed by change in plasma norepinephrine. | 2 weeks
The effects of a 2-week trial of nasal oxytocin compared with placebo on maternal reactivity to a social stressor indexed by self-reported affective ratings. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Grewen, Ph.D., Principal Investigator — UNC School of Medicine, Dept. of Psychiatry
Locations (1):
- UNC School of Medicine, Medical School Wing D, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No